CLINICAL TRIAL: NCT06789133
Title: Effects of Gait Training With and Without Proprioceptive Neuromuscular Facilitation on Balance, Gait and Activities of Daily Living in Parkinson's Patients
Brief Title: Effects of Gait Training With and Without PNF on Balance ,Gait and Activities of Daily Living in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0215KainatAhmad
Record Dates: First submitted 2024-12-20; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease (PD); Proprioceptive Neuromuscular Facilitation
Keywords: PNF; PD; BWSTT; ADLs
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF exercises and Body weight supported treadmill gait training (Experimental): PNF exercises and Body weight supported treadmill gait training
  Interventions: Other: PNF exercises and Body weight supported treadmill gait training
- Gait training without PNF (Active Comparator): Treadmil gait training and Routine physical therapy
  Interventions: Other: Body weight supported treadmill gait training and Routine physical therapy

INTERVENTIONS:
Other: PNF exercises and Body weight supported treadmill gait training — PNF Exercises:
  .Proprioceptive neuromuscular facilitation exercises include D1 Flexion and D1 Extension of lower limb ,D2 flexion D2 extension of lower limb .rhythmic initiation ,hold relax ,pelvic pattern and contract relax technique . subjects will perform each exercise for 30sec with resting interval of 30 to 60 seconds Will be provided after completion of each exercise. 3 sessions will be held per week, For 8 weeks
  Gait training:
  Body weight supported treadmill gait training for 20 minutes 3 sessions per week.
  In total all PNF exercises with gait training will be held for 40-45 minutes.
  Arms: PNF exercises and Body weight supported treadmill gait training
Other: Body weight supported treadmill gait training and Routine physical therapy — Body Weight Supported Treadmill Training (BWSTT):
  This will include body weight supported treadmill gait training. 10 % BWSTT or 20% BWSTT. The session will of 20 minutes .3 sessions will be Held per week.
  Routine physical therapy:
  Stretching and strengthening of lower extremities In total all BWSTT along with routine physical therapy protocol will be held for 40-45minutes .3 sessions will be held per week.
  Arms: Gait training without PNF

SUMMARY:
Proprioceptive Neuromuscular Facilitation (PNF) and gait training exercises are specifically used to treat balance, gait and functional activities in Parkinson s patients. PNF has been compared with gait training and balance training in other conditions like stroke and multiple sclerosis but limited literatures are present in which PNF has been compared with gait training in Parkinson patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's patients.
* Patients from both gender around the age of 45-65.
* Patient with a score of 42 above on the Berg Balance Scale.
* Patients with shuffling gait
* Patient with good cognitive function minimum score of 20 or more on Mini-mental Status Examination MMSE scale
* Exclusion Criteria:
* Patients with a history of CVA.
* Patient with peripheral vascular disease.
* Patient with fracture or dislocation of lower limb.
* Patient with peripheral nerve injury

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 4 weeks
  The Berg Balance Scale (BBS) is a test that measures a person's balance abilities by asking them to perform 14 simple tasks, such as standing, sitting, reaching, and turning. The test is scored on a scale from 0 to 56, with higher scores indicating better balance. The BBS is used to assess people who have balance impairments due to various conditions, such as stroke, Parkinson's disease, osteoarthritis, or inner ear problems. The BBS has been shown to have good reliability and validity for measuring balance in Ho The reliability and validity of this test is 0.95 or 95%
Time up and go Test | 4 weeks
  from baseline :The Time Up and Go (TUG) test is a simple and quick test that measures a person's functional mobility and fall risk. The test involves standing up from a chair, walking 10 feet, turning around, walking back, and sitting down again, while timing how long it takes to complete the task. The TUG test is used to evaluate people who have balance impairments due to various conditions, such as aging, stroke, Parkinson's disease, or vestibular disorders. The TUG test also has some limitations. The reliability of this test is 0.97 to o.99.
Modified Barthel index | 4 weeks
  The Barthel Index is a scale used to measure an individual's ability to perform activities of daily living. The Reliability of MBI is 0.73 to 0.77. It is often employed in healthcare settings to evaluate functional independence, guide rehabilitation plans, and monitor progress in patients. there are 10 items, each scored from 0 to 2 or 3 points, The total score ranges from 0 to 20 or 25, with higher scores indicating greater independence. The 10 items are:
  Bowel control Bladder control Grooming Toilet using Feeding Transfer (bed to chair and back) Mobility Dressing Stairs Bathing

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, MSDPT, Principal Investigator — Riphah International University
Locations (1):
- Arthritis and spine care , Lahore General hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazhar T, Jameel A, Sharif F, Asghar M. Effects of conventional physical therapy with and without proprioceptive neuromuscular facilitation on balance, gait, and function in patients with Parkinson's disease. J Pak Med Assoc. 2023 Jun;73(6):1280-1283. doi: 10.47391/JPMA.6710. PMID 37427630
- [Background] Giardini M, Nardone A, Godi M, Guglielmetti S, Arcolin I, Pisano F, Schieppati M. Instrumental or Physical-Exercise Rehabilitation of Balance Improves Both Balance and Gait in Parkinson's Disease. Neural Plast. 2018 Mar 7;2018:5614242. doi: 10.1155/2018/5614242. eCollection 2018. PMID 29706993
- [Background] Alexandre de Assis IS, Luvizutto GJ, Bruno ACM, Sande de Souza LAP. The Proprioceptive Neuromuscular Facilitation Concept in Parkinson Disease: A Systematic Review and Meta-Analysis. J Chiropr Med. 2020 Sep;19(3):181-187. doi: 10.1016/j.jcm.2020.07.003. Epub 2020 Dec 15. PMID 33362441
- [Background] Mak MKY, Wong-Yu ISK. Exercise for Parkinson's disease. Int Rev Neurobiol. 2019;147:1-44. doi: 10.1016/bs.irn.2019.06.001. Epub 2019 Jun 27. PMID 31607351
- [Background] Pelicioni PHS, Menant JC, Latt MD, Lord SR. Falls in Parkinson's Disease Subtypes: Risk Factors, Locations and Circumstances. Int J Environ Res Public Health. 2019 Jun 23;16(12):2216. doi: 10.3390/ijerph16122216. PMID 31234571
- [Background] Mirelman A, Bonato P, Camicioli R, Ellis TD, Giladi N, Hamilton JL, Hass CJ, Hausdorff JM, Pelosin E, Almeida QJ. Gait impairments in Parkinson's disease. Lancet Neurol. 2019 Jul;18(7):697-708. doi: 10.1016/S1474-4422(19)30044-4. Epub 2019 Apr 8. PMID 30975519
- [Background] Nonnekes J, Nieuwboer A. Towards Personalized Rehabilitation for Gait Impairments in Parkinson's Disease. J Parkinsons Dis. 2018;8(s1):S101-S106. doi: 10.3233/JPD-181464. PMID 30584154